CLINICAL TRIAL: NCT03605433
Title: Surgical Coronary Revascularization Outcomes After Oral Anticoagulation or Antiplatelet Strategies
Brief Title: Surgical Revascularization Outcomes After Oral Anticoagulation or Antiplatelets
Acronym: SCOOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Luís Paiva, Luis Paiva, Unidade Local de Saúde de Coimbra, EPE
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCOOP
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease; Saphenous Vein Graft Patency
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Anticoagulation+Antiplatelet (Experimental): Rivaroxaban 2.5 mg twice daily and Aspirin 100 mg once daily.
  Interventions: Drug: Rivaroxaban
- Oral Anticoagulation (Experimental): Rivaroxaban 20 mg once daily
  Interventions: Drug: Rivaroxaban
- Antiplatet (Active Comparator): Aspirin 100 mg once daily
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 2.5 mg or Rivaroxaban 20 mg or no oral anticoagulation

SUMMARY:
The primary purpose of this study is to evaluate whether treatment with oral anticoagulation or oral anticoagulation and aspirin is better than aspirin alone in cardiovascular outcomes and saphenous graft patency in patients submitted to coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to coronary artery bypass graft and at least one saphenous vein graft

Exclusion Criteria:

* Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy or oral anticoagulant therapy
* Stroke within 1 month or any history of hemorrhagic or lacunar stroke
* Estimated glomerular filtration rate (eGFR)<15 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 5 years
  Time from randomization to the first occurrence of either myocardial infarction, stroke, or cardiovascular death
Graft Patency | 5 years
  Time from randomization to the first occurence of saphenous graft oclusion
Major Bleeding | 5 years
  Time from randomization to the first occurrence of major bleeding (modified International Society on Thrombosis and Haemostasis)

SECONDARY OUTCOMES:
MACE, cardiovascular death | 5 years
  Time from randomization to first occurrence of either coronary heart disease death, myocardial infarction, ischemic stroke, acute limb ischemia
All-cause mortality | 5 years
  Time from randomization to first occurrence of all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided